CLINICAL TRIAL: NCT03830671
Title: The Effect of New MDR-TB Regimen With 18 Month Duration Containing 6 Anti-tuberculosis Drugs
Brief Title: The Effect of 18-month Regimen Containing 6 Anti-tuberculosis Drugs for Patients With MDR-TB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Qi Li, Director of Tuberculosis Clinical Research, Beijing Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018ZX10722301-001
Record Dates: First submitted 2019-01-31; First posted 2019-02-05 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Multi-drug Resistant Tuberculosis
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- investigational arm (Experimental): the arm was given investigational regimen:3Am-Mfx-PZA-X-Y-Z/3Am3-Mfx-PZA-X-Y-Z/12 Mfx-PZA-X-Y-Z.X、Y、Z are the drugs susceptible or possibly susceptible to mycobacterial bacilli(The candidated drugs to be selected are:Cs-Cycloserine,Pto-Protionamide,Clr-Clarithromycin,PAS-sodium para-aminosalicylate,E-ethambutol,Bdq-Bedaquiline,Cfz-Clofazimine,Lzd-linezolid).The abbreviation of the name of each drug in the regimen is explained as follows: PZA-pyrazinamide，Am-Amikacin，Mfx-moxifloxacin）and the total duration of the regimen is 18 months.
  Interventions: Drug: 18-month regimen containing 6 anti-TB drugs

INTERVENTIONS:
Drug: 18-month regimen containing 6 anti-TB drugs — Investigational regimen:3Am-Mfx-PZA-X-Y-Z/3Am3-Mfx-PZA-X-Y-Z/12 Mfx-PZA-X-Y-Z.X、Y、Z are the drugs susceptible or possibly susceptible to mycobacterial bacilli(The candidated drugs to be selected are:Cs-Cycloserine,Pto-Protionamide,Clr-Clarithromycin,PAS-sodium para-aminosalicylate,E-ethambutol,Bdq-Bedaquiline,Cfz-Clofazimine,Lzd-linezolid).The abbreviation of the name of each drug in the regimen is explained as follows: PZA-pyrazinamide，Am-Amikacin，Mfx-moxifloxacin）and the total duration of the regimen is 18 months

SUMMARY:
WHO has recommended that multidrug-resistant tuberculosis (MDR-TB, defined as resistance to at least isoniazid (H) and rifampicin (R) be addressed as a public health crisis and enhance capacity to deliver effective treatment and care. According to the 2018 WHO TB Report, the overall treatment success rate of MDR-TB is 55% while much lower in China at just only 41% with the 24-month regimen. In order to further verify the safety and efficiency of optimizing shorter 18-month regimen containing 6 anti-TB drugs with MDR-TB patients,500 more patients will be enrolled and observed.

DETAILED DESCRIPTION:
1. Design: the study is a multi-center,open, single arm trial.
2. Population:patients with sputum culture positive and confirmed as MDR-TB via drug resistance of isoniazid(H),rifampicin(R),ethambutol(E)and pyrazinamide or patients with GeneXpert confirmed RR-TB.
3. Investigational regimen:3Am-Mfx-PZA-X-Y-Z/3Am3-Mfx-PZA-X-Y-Z/12 Mfx-PZA-X-Y-Z.X、Y、Z are the drugs susceptible or possibly susceptible to mycobacterial bacilli(The candidated drugs to be selected are:Cs-Cycloserine,Pto-Protionamide,Clr-Clarithromycin,PAS-sodium para-aminosalicylate,E-ethambutol,Bdq-Bedaquiline,Cfz-Clofazimine,Lzd-linezolid).The abbreviation of the name of the 3 drugs in the regimen is explained as follows: PZA-pyrazinamide，Am-Amikacin，Mfx-moxifloxacin）and the total duration of the regimen is 18 months.
4. Primary and secondary outcome measures:

   The primary outcome measures include 1.the treatment success rate.2. Death rate.

   The secondary outcome measures include 1.sputum conversion rate at the end of month 2, month 3,intensive phase of 6 months and treatment completion of all enrolled patients.2.Frequency of adverse drug reaction occurring during treatment.3.Radiological manifestation change of TB lesion or cavity during treatment.
5. Sample size: 500 eligible patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to give informed consent to participate in the trial treatment and follow-up.
* Is aged between 18 years and 70 years.
* Has a positive sputum culture result or a positive GeneXpert result.
* Has evidence of RR-TB or MDR-TB either by GeneXpert or culture-based drug susceptibility testing (DST).
* Non pre-XDR-TB or XDR-TB.
* Is willing to use effective contraception of women at childbearing age.
* Has had a chest X-ray that is compatible with a diagnosis of pulmonary TB.

Exclusion Criteria:

* pre-XDR-TB or XDR-TB.
* Has a known allergy to any drug of the regimen.
* Is currently taking or took part in another trial less than three months before the study initiation .
* Is HIV positive.
* Has abnormal ECG with QT prolongation over 430ms of men while 450 of women.
* Is critically ill, and in the judgment of the investigator, unlikely to take part in the study.Or has any condition (social or medical) which in the opinion of the investigator would make study participation unsafe.
* Is known to be pregnant or breast-feeding.
* Has severe cardiovascular diseases, such as heart failure, hypertension (poor blood pressure control), arrhythmia or post-infarction status.
* Has severe concomitant severe disease such as respiratory failure or cardiac insufficiency or liver and kidney injury with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 2.5 times the upper limit of normal or with serum creatinine(Cr)more than 1.3 times the upper limit of normal.
* Has Karnofsky score less than 50%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
the treatment success rate | at the end of treatment completion of all enrolled patients,an average of 18 months after the last patient enrolled
death rate | at the end of treatment completion of all enrolled patients, an average of 18 months after the last patient enrolled

SECONDARY OUTCOMES:
sputum conversion rate at the end of month 2, month 3,intensive phase and treatment completion. | at the end of month 2, month 3,intensive phase of 6 months since treatment initiation and treatment completion of all enrolled patients, an average of 18 months after the last enrolled patient.
Frequency of adverse drug reaction occurring during treatment. | at the end of treatment completion of all enrolled patients, an average of 18 months after the last enrolled patient.
Radiological manifestation change of TB lesion or cavity at the end of month 2, month 3,intensive phase and treatment completion. | at the end of month 2, month 3,intensive phase of 6 months since treatment initiation and treatment completion of all enrolled patients, an average of 18 months after the last enrolled patient.
  proportion of lung field the lesion accumulated taken up at different time points with the comparison to that at baseline. The number and size of cavities at different time points with comparison to that at baseline.

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Beijing Chest Hospital, Beijing
  - The 8th Medical Center of Chinese Pla General Hospital, Beijing
  - Changchun Infectious Disease Hospital, Changchun
  - Hunan Institute For Tuberculosis Control, Changsha
  - Public Health Clinical Center of Chengdu, Chengdu
  - Shenzhen Third Peple's Hospital, Guangzhou
  - Guangzhou Chest Hospital, Guanzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Infectious Disease Prevention Hospital in Heilongjiang Province, Harbin
  - Anhui Chest Hospital, Hefei
  - The Fourth People's Hospital of Inner Mongolia Autonomous region, Hohhot
  - Shandong Provincial Chest Hospital, Jinan
  - Shanghai Pulmonary Hospital, Shanghai
  - Shenyang Chest Hospital, Shenyang
  - Tianjin Haihe Hospital, Tianjin
  - Chest of Hospital of Xinjiang Uygur Autonomous Region of the PRC, Ürümqi
  - The Tuberculosis Prevention and Treatment Hospital of Shanxi Province, Xi'an
  - Xi'an Chest Hospital, Xi'an
  - The Fourth People's Hospital of Ningxia Autonomous Region, Yinchuan
  - The Infectious Disease Hospital of Wangkai Zaozhuang, Zaozhuang